CLINICAL TRIAL: NCT01903460
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of LUM001, an Apical Sodium-dependent Bile Acid Transporter Inhibitor (ASBTi), in the Treatment of Cholestatic Liver Disease in Paediatric Patients With Alagille Syndrome
Brief Title: Safety and Efficacy Study of LUM001 in the Treatment of Cholestatic Liver Disease in Patients With Alagille Syndrome
Acronym: IMAGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUM001-302; 2012-005346-38 (EudraCT Number); SHP625-302 (Other: Shire Development LLC)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LUM001 (Experimental): LUM001 administered orally once each day
  Interventions: Drug: LUM001
- Placebo (Placebo Comparator): Placebo administered orally once each day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LUM001
  Arms: LUM001
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of LUM001. Efficacy will be assessed by evaluating the effect of LUM001 versus placebo on the biochemical markers and pruritus associated with Alagille Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Alagille Syndrome
2. Evidence of cholestasis
3. Moderate to severe pruritus
4. Ability to understand and willingness to sign informed consent/assent prior to initiation of any study procedures

Exclusion Criteria:

1. Surgical disruption of the enterohepatic circulation
2. Liver transplant
3. History or presence of other concomitant liver disease
4. Females who are pregnant or lactating
5. Known HIV infection

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (3):
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham, West Midlands
  - Leeds Teaching Hospitals, Leeds, West Yorkshire
  - Kings College Hospital, London

RESULTS

PARTICIPANT FLOW:
Groups:
- LUM001 140ug/kg/Day: Participants received an escalating dose of LUM001 over 3 to 5 weeks, from 14ug/kg/day to 140ug/kg/day, then received 8 to 10 weeks of treatment at either 140ug/kg/day or the highest tolerated dose below 140ug/kg/day. Participants were then followed for 4 weeks after treatment.
- LUM001 280ug/kg/Day: Participants received an escalating dose of LUM001 over 3 to 5 weeks, from 14ug/kg/day to 280ug/kg/day, then received 8 to 10 weeks of treatment at either 280ug/kg/day or the highest tolerated dose below 280ug/kg/day. Participants were then followed for 4 weeks after treatment.
- Placebo Cohort A; Placebo Cohort B: Participants received LUM001-matching placebo for up to 13 weeks, then were followed for 4 weeks after treatment.
Period: Overall Study
Arm/Group | LUM001 140ug/kg/Day | LUM001 280ug/kg/Day | Placebo Cohort A | Placebo Cohort B
Started | 6 | 8 | 3 | 3
Completed | 6 | 8 | 3 | 2
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | LUM001 140ug/kg/Day | LUM001 280ug/kg/Day | Placebo Cohort A | Placebo Cohort B | Total
Number analyzed (Participants) | 6 | 8 | 3 | 3 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (4.49) | 6.8 (6.73) | 5.0 (2.00) | 4.3 (3.21) | 5.9 (4.93)
Age, Customized [Number; unit: participants]
  < 2 years | 0 | 3 | 0 | 0 | 3
  2 to 4 years | 3 | 1 | 1 | 2 | 7
  5 to 8 years | 1 | 1 | 2 | 1 | 5
  9 to 12 years | 2 | 0 | 0 | 0 | 2
  13 to 18 years | 0 | 3 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 2 | 10
  Male | 4 | 5 | 0 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 8 | 3 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 (End of Treatment) in Fasting Serum Bile Acid Level
Description: Participants were required to fast for at least 4 hours; only water was permitted prior to collection. A negative change from baseline indicates that the level of bile acid decreased.
Time Frame: Baseline to 13 weeks or end of treatment
Population: The modified Intent-to-Treat (mITT) population, defined as all participants in the Safety population who had at least 1 post-baseline efficacy assessment. The Safety population was defined as all participants who were randomly assigned to study treatment and who received any amount of study drug.
Measure: Least Squares Mean (Standard Error); unit: umol/L
Groups:
- LUM001 Overall: Participants received either dose of LUM001 for up to 10 or 13 weeks, then were followed for 4 weeks after treatment.
- Placebo Overall: Participants received LUM001-matching placebo for up to 13 weeks, then were followed for 4 weeks after treatment.
Arm/Group | LUM001 140ug/kg/Day | LUM001 280ug/kg/Day | LUM001 Overall | Placebo Overall
Number analyzed (Participants) | 6 | 8 | 14 | 6
umol/L | -82.864 (50.1513) | -49.388 (43.4732) | -66.126 (33.1208) | -42.157 (50.0903)
Statistical Analysis 1: Comparison: LUM001 140ug/kg/Day vs Placebo Overall; Analysis of LUM001 140ug/kg/day; Test type: Superiority or Other; p = 0.5740, ANCOVA; LS mean difference from placebo = -40.707, 95% CI 2-sided [-191.679 to 110.265]
Statistical Analysis 2: Comparison: LUM001 280ug/kg/Day vs Placebo Overall; Analysis of LUM001 280ug/kg/day; Test type: Superiority or Other; p = 0.9147, ANCOVA; LS mean difference from placebo = -7.231, 95% CI 2-sided [-148.726 to 134.264]
Statistical Analysis 3: Comparison: LUM001 Overall vs Placebo Overall; Analysis of all doses of LUM001; Test type: Superiority or Other; p = 0.6954, ANCOVA; LS mean difference from placebo = -23.969, 95% CI 2-sided [-151.969 to 104.031]

2. Secondary Outcome: Change From Baseline to Week 13 (End of Treatment) in Liver Enzymes
Description: Analysis of liver enzymes included alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP). A negative change from baseline indicates that the level of that enzyme decreased.
Time Frame: Baseline to 13 weeks or end of treatment
Population: The mITT population, defined as all participants in the Safety population who had at least 1 post-baseline efficacy assessment. The Safety population was defined as all participants who were randomly assigned to study treatment and who received any amount of study drug.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | LUM001 140ug/kg/Day | LUM001 280ug/kg/Day | LUM001 Overall | Placebo Overall
Number analyzed (Participants) | 6 | 8 | 14 | 6
U/L
  ALT | 59.3 (20.99) | 10.5 (18.06) | 34.9 (13.86) | 2.7 (21.06)
  AST | 37.2 (13.64) | -2.7 (11.70) | 17.3 (8.98) | 13.2 (13.63)
  ALP | 71.4 (53.35) | 31.6 (43.59) | 51.5 (36.13) | 19.7 (60.76)
Statistical Analysis 1: Comparison: LUM001 140ug/kg/Day vs Placebo Overall; Analysis of LUM001 140ug/kg/day for ALT; Test type: Superiority or Other; p = 0.0783, ANCOVA; LS mean difference from placebo = 56.7, 95% CI 2-sided [-7.2 to 120.6]
Statistical Analysis 2: Comparison: LUM001 280ug/kg/Day vs Placebo Overall; Analysis of LUM001 280ug/kg/day for ALT; Test type: Superiority or Other; p = 0.7827, ANCOVA; LS mean difference from placebo = 7.8, 95% CI 2-sided [-51.4 to 67.0]
Statistical Analysis 3: Comparison: LUM001 Overall vs Placebo Overall; Analysis of all doses of LUM001 for ALT; Test type: Superiority or Other; p = 0.2235, ANCOVA; LS mean difference from placebo = 32.2, 95% CI 2-sided [-21.9 to 86.3]
Statistical Analysis 4: Comparison: LUM001 140ug/kg/Day vs Placebo Overall; Analysis of LUM001 140ug/kg/day for AST; Test type: Superiority or Other; p = 0.2372, ANCOVA; LS mean difference from placebo = 24.0, 95% CI 2-sided [-17.5 to 65.5]
Statistical Analysis 5: Comparison: LUM001 280ug/kg/Day vs Placebo Overall; Analysis of LUM001 280ug/kg/day for AST; Test type: Superiority or Other; p = 0.3914, ANCOVA; LS mean difference from placebo = -15.8, 95% CI 2-sided [-54.1 to 22.4]
Statistical Analysis 6: Comparison: LUM001 Overall vs Placebo Overall; Analysis of all doses of LUM001 for AST; Test type: Superiority or Other; p = 0.8081, ANCOVA; LS mean difference from placebo = 4.1, 95% CI 2-sided [-31.0 to 39.1]
Statistical Analysis 7: Comparison: LUM001 140ug/kg/Day vs Placebo Overall; Analysis of LUM001 140ug/kg/day for ALP; Test type: Superiority or Other; p = 0.5748, ANCOVA; LS mean difference from placebo = 51.7, 95% CI 2-sided [-140.3 to 243.7]
Statistical Analysis 8: Comparison: LUM001 280ug/kg/Day vs Placebo Overall; Analysis of LUM001 280ug/kg/day for ALP; Test type: Superiority or Other; p = 0.8835, ANCOVA; LS mean difference from placebo = 11.9, 95% CI 2-sided [-158.4 to 182.2]
Statistical Analysis 9: Comparison: LUM001 Overall vs Placebo Overall; Analysis of all doses of LUM001 for ALP; Test type: Superiority or Other; p = 0.6917, ANCOVA; LS mean difference from placebo = 31.8, 95% CI 2-sided [-135.8 to 199.4]

3. Secondary Outcome: Change From Baseline to Week 13 (End of Treatment) in Pruritus as Measured by The Patient And Observer Itch Reported Outcome (ItchRO) Average Daily Scores
Description: The ItchRO was administered as a twice daily electronic diary (eDiary). Children ≥9 years of age completed the patient ItchRO; those between the ages of 5 and 8 completed the patient ItchRO with the assistance of their caregiver. There was no patient report for subjects under the age of 5. ItchRO scores range from 0 to 4, with the higher score indicating increasing itch severity. ItchRO average daily scores were calculated as the sum of daily scores (ie, the maximum of morning and evening scores) divided by the number of days. The average daily score was calculated by using the 7 days pre-treatment for baseline, and the last 7 days of treatment for Week 13. A negative change from Baseline indicates that itch severity decreased.
Time Frame: Baseline to 13 weeks or end of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LUM001 140ug/kg/Day | LUM001 280ug/kg/Day | LUM001 Overall | Placebo Overall
Number analyzed (Participants) | 6 | 8 | 14 | 6
units on a scale
  Patient ItchRO | -1.159 (0.5396) | -0.608 (0.4399) | -0.883 (0.3484) | -0.811 (0.5684)
  Observer ItchRO | -0.802 (0.2732) | -0.419 (0.2318) | -0.610 (0.1776) | -0.592 (0.2690)
Statistical Analysis 1: Comparison: LUM001 140ug/kg/Day vs Placebo Overall; Analysis of LUM001 140ug/kg/day for Patient ItchRO; Test type: Superiority or Other; p = 0.6907, ANCOVA; LS mean difference from placebo = -0.348, 95% CI 2-sided [-2.468 to 1.772]
Statistical Analysis 2: Comparison: LUM001 280ug/kg/Day vs Placebo Overall; Analysis of LUM001 280ug/kg/day for Patient ItchRO; Test type: Superiority or Other; p = 0.7897, ANCOVA; LS mean difference from placebo = 0.202, 95% CI 2-sided [-1.647 to 2.052]
Statistical Analysis 3: Comparison: LUM001 Overall vs Placebo Overall; Analysis of all doses of LUM001 for Patient ItchRO; Test type: Superiority or Other; p = 0.9203, ANCOVA; LS mean difference from placebo = -0.073, 95% CI 2-sided [-1.850 to 1.705]
Statistical Analysis 4: Comparison: LUM001 140ug/kg/Day vs Placebo Overall; Analysis of LUM001 140ug/kg/day for Observer ItchRO; Test type: Superiority or Other; p = 0.5966, ANCOVA; LS mean difference from placebo = -0.210, 95% CI 2-sided [-1.038 to 0.618]
Statistical Analysis 5: Comparison: LUM001 280ug/kg/Day vs Placebo Overall; Analysis of LUM001 280ug/kg/day for Observer ItchRO; Test type: Superiority or Other; p = 0.6320, ANCOVA; LS mean difference from placebo = 0.173, 95% CI 2-sided [-0.580 to 0.926]
Statistical Analysis 6: Comparison: LUM001 Overall vs Placebo Overall; Analysis of all doses of LUM001 for Observer ItchRO; Test type: Superiority or Other; p = 0.9547, ANCOVA; LS mean difference from placebo = -0.019, 95% CI 2-sided [-0.710 to 0.673]

ADVERSE EVENTS:
Arm/Group | LUM001 140ug/kg/Day | LUM001 280ug/kg/Day | Placebo Overall
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 7/8 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LUM001 140ug/kg/Day (N=6) | LUM001 280ug/kg/Day (N=8) | Placebo Overall (N=6)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (8) | 1 (5)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (4) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 5 (9) | 2 (3)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Crying (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (2) | 3 (6)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually